CLINICAL TRIAL: NCT06205225
Title: iCardia4HF: A Multi-component mHealth App and Tailored Text-messaging Intervention to Promote Self-care Adherence and Improve Health Outcomes in Patients With Chronic Heart Failure
Brief Title: iCardia4HF: Multi-component mHealth Intervention for Patients With Heart Failure
Acronym: iCardia4HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Spyros Kitsiou, Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-1592; R01HL168376 (NIH)
Record Dates: First submitted 2024-01-03; First posted 2024-01-12 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure
Keywords: mHealth, wearables, mobile apps, heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: 2 x 2 factorial randomized controlled trial
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Care providers who provide usual care to study participants will be unaware of the study groups and group assignments. Outcome assessors will be masked to group assignment. Outcome assessors will work in a different office from other study investigators and will have limited access to the Electronic Data Capturing system used for data collection (REDCap).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Enhanced usual care (Active Comparator): Participants assigned to the usual care group will receive (1) standard care, (2) patient education about HF self-care, and (3) three connected health devices. Usual care includes follow-up appointments every 2-3 months with a multidisciplinary team at the outpatient HF clinic. Patient education includes resources about HF self-care from the American Heart Association and Heart Failure Society of America. Connected health devices include the Withings Weight Scale, Withings blood pressure monitor, and Fitbit Charge 6 activity tracker (wrist-based with heart rate sensor). Participants will receive the devices at baseline along with training by research staff on how to use the devices to perform daily self-monitoring of weight, blood pressure, and physical activity/inactivity. The Withings devices have a cellular antenna for automatic transmission of data to our study server (iCardia). Fitbit will be paired with the participant's smartphone.
  Interventions: Behavioral: Enhanced Usual Care
- Text4HF (Experimental): Participants allocated to the Text4HF group will receive the same components and devices as the usual care group (usual care, patient education, and connected health devices), plus individually tailored Text Messages targeting health beliefs, HF-knowledge, and self-efficacy about HF self-care. Participants will receive 4-6 TMs/week during the induction phase (0 to 3 months), and 2-4 TMs per week during the adoption period (3 to 6 months).Tailoring of the TMs is guided by participants' responses to validated instruments assessing intervention target variables at baseline and 3 months
  Interventions: Behavioral: Text4HF
- MyApps (Experimental): In addition to usual care and patient education resources, participants in the MyApps group will receive three commercially available apps (Heart Failure Storylines, Withings Health Mate, and Fitbit), and three connected health devices (Withings Body Cardio Scale, Withings BP monitor, and Fitbit activity tracker). The apps interface with the devices via Bluetooth offering patients a comprehensive set of mHealth tools that support the core elements of HF self-care (maintenance, self-monitoring, and self-management).
  Interventions: Behavioral: MyApps
- MyApps + Text4HF (Experimental): Participants in this group will receive the MyApps and Text4HF intervention components, combined.
  Interventions: Behavioral: MyApps & Text4HF

INTERVENTIONS:
Behavioral: Text4HF — Behavioral text messages about heart failure self-care
  Arms: Text4HF
Behavioral: MyApps — consumer mobile health apps and devices for heart failure self-care
  Arms: MyApps
Behavioral: MyApps & Text4HF — Consumer mobile health apps and devices supplemented with behavioral text messages for heart failure self-care
  Arms: MyApps + Text4HF
Behavioral: Enhanced Usual Care — Participants assigned to the enhanced usual care group will receive (1) standard care, (2) patient education about HF self-care, and (3) three connected health devices (Withings weight scale and blood pressure monitor, and Fitbit activity tracker with Fitbit mobile app).
  Arms: Enhanced usual care

SUMMARY:
The goal of this factorial randomized trial is to examine the independent and synergistic efficacies of two mobile health technology interventions in people with chronic heart failure. The first intervention involves the use of multiple consumer mHealth apps and sensor devices (MyApps) for heart failure self-care (maintenance, monitoring, and management). The second intervention is a program of tailored text messages (Text4HF) targeting modifiable behavioral factors associated with heart failure self-care non-adherence. The main questions this study aims to answer are:

1. Can the use of consumer mHealth apps and devices (MyApps) improve heart failure self-care and reduce days lost due to cardiovascular hospitalization or death for any cause?
2. Can a program of individually tailored text messages (Text4HF) improve heart failure self-care and reduce the days lost due to cardiovascular hospitalization or death for any cause?
3. Can MyApps and Text4HF combined lead to greater improvements in heart failure self-care and days lost due to cardiovascular hospitalization or death for any cause

DETAILED DESCRIPTION:
Heart failure (HF) remains one of the most frequent principal diagnoses for hospitalization and a leading cause of death in the United States. Up to 65% of HF readmissions are the result of insufficient self-care. Existing HF self-care interventions delivered face-to-face or via telephone have had limited impact and reach. They require significant provider time and are not always accessible to patients. There is an urgent need for accessible and scalable interventions that are designed to assist patients with HF self-care while in the community to reduce HF readmissions. Consumer mobile health (mHealth) technologies (e.g., mobile apps and sensor devices) hold promise for promoting HF self-care and expanding intervention delivery. However, their efficacy remains largely underexplored.

To address this gap, our team developed a patient-centered HF self-care intervention (iCardia4HF) that combines the use of three consumer mobile health apps and connected health devices (MyApps) with a program of individually tailored text messages (Text4HF) targeting modifiable behavioral factors to promote HF self-care adherence and improve clinical outcomes.

This study aims to conduct a fully powered, 2x2 factorial randomized controlled trial to determine the independent and combined efficacy of the two iCardia4HF intervention components (MyApps and Text4HF) at 6 months, as well as their maintenance efficacy at 6 months post-intervention. A total of 360 patients with HF will be recruited and randomized to one of four conditions for 12 months: (1) Usual care, (2) Text4HF, (3) MyApps, or (4) MyApps&Text4HF. Specific aims are:

Aim 1: Determine the independent and combined efficacies of MyApps and Text4HF at 6-months on the primary outcome of days lost due to cardiovascular hospitalization or death for any cause, and secondary outcomes of HF self-care and health status.

Hypothesis 1a: MyApps and Text4HF will have significant main effects on the primary outcome at 6 months.

Hypothesis 1b: MyApps and Text4HF will have significant main effects on objectively assessed measures of HF self-care adherence, self-reported HF self-care, and health status, at 6 months.

Aim 2: Determine the independent and combined maintenance efficacies of MyApps and Text4HF at 12 months (6 months post-intervention).

Hypothesis 2a: Text4HF and MyApps will have significant main effects on the primary outcome at 12 months.

Hypothesis 2b: Text4HF and MyApps will have significant main effects on objectively assessed measures of HF self-care adherence, self-reported HF self-care, and health status, at 12 months.

Aim 3: Investigate the mediating effect of intervention targets (health beliefs, HF knowledge, self-efficacy), and moderating effect of multi-level determinants of HF self-care adherence on the efficacy of the intervention, across individual (e.g., age, race/ethnicity), illness-related (e.g., depression, comorbidities), and socioeconomic factors (e.g., insurance, income, employment, and access to care).

Impact statement: This study will provide important new knowledge that will critically shape our understanding about the potential of commercially available mHealth technologies and tailored text messages to improve HF self-care adherence and reduce hospital readmissions in patients with HF.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Stage C Heart Failure
* ≥ 18 years of age
* Transthoracic Echocardiogram or Cardiac MRI performed in the last 3 years and LVEF results available
* Patient is actively treated with oral loop diuretics for chronic heart failure
* Hospitalization due to acute decompensated heart failure within 24 months before randomization and/or insufficient self-care per SCHFI assessment (score of ≤3, in at least two items of the SCHFI v7.2 maintenance, symptom monitoring, or self-care management subscale)
* Ability to speak and read English

Exclusion Criteria:

* Implanted ventricular assist device
* High urgent listed for heart transplantation
* Acute coronary syndrome within the last 7 days before randomization
* Revascularization and/or CRT implantation within 28 days before randomization
* Planned revascularization, transcatheter aortic valve implantation, MitraClip and/or CRT implantation within 3 months after randomization
* End-stage HF (hospice candidate)
* Discharge to a setting other than home
* Individuals who have a home nurse or are not able to take care of self (eat, dress, walk, bathe, take medications, or use the toilet)
* Chronic renal insufficiency with hemodialysis or estimated Glomerular Filtration Rate <25 mL
* Active cancer, currently undergoing treatment (e.g. radiation immunotherapy)
* Existence of any disease reducing life expectancy to less than 1 year
* Cognitive impairment (e.g., Dementia, Parkinson disease, Alzheimer disease, MoCA<18, impaired self-determination, lacking ability to communicate)
* Major physical impairment (e.g., inability to walk, bound on a wheelchair)
* Unwillingness to use study equipment
* Active substance abuse
* Currently pregnant, less than 3-month post-partum or pregnancy anticipated during the study
* Participation in other treatment studies or remote patient management programs
* Participation in the iCardia4H pilot trial (conducted before this study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-10-04 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of days lost due to unplanned cardiovascular hospitalizations or death from any cause | 6 months
  Hospitalization is defined as hospital admission resulting in an overnight stay where the length of stay is at least 24 hours. Events leading to emergency department visit only with a length of stay under 24 hours will not be classified as hospitalization. For a hospitalization to be considered as unplanned the patient must present new symptoms and/or worsening of existing symptoms with the need for immediate admission in a hospital for intensified care. A hospitalization will be considered "cardiovascular" when it is due to cardiovascular causes which includes but is not limited to: HF deterioration, acute myocardial infarction, arrhythmia, HF, pulmonary embolism, cerebrovascular disease (e.g., stroke), severe bleeding, endocarditis, etc.

SECONDARY OUTCOMES:
Percentage of days lost due to unplanned cardiovascular hospitalizations or death from any cause | 12 months
  Hospitalization is defined as hospital admission resulting in an overnight stay where the length of stay is at least 24 hours. Events leading to emergency department visit only with a length of stay under 24 hours will not be classified as hospitalization. For a hospitalization to be considered as unplanned the patient must present new symptoms and/or worsening of existing symptoms with the need for immediate admission in a hospital for intensified care. A hospitalization will be considered "cardiovascular" when it is due to cardiovascular causes which includes but is not limited to: HF deterioration, acute myocardial infarction, arrhythmia, HF, pulmonary embolism, cerebrovascular disease (e.g., stroke), severe bleeding, endocarditis, etc.
Number of patients with unplanned cardiovascular hospitalizations | 6 and 12 months
  Number of patients with one or more unplanned cardiovascular-related hospitalizations
Mean number of unplanned cardiovascular hospitalizations | 6 and 12 months
  Mean number of unplanned hospital admissions for cardiovascular reasons
Unplanned heart failure hospitalizations | 6 and 12 months
  Number of patients with one or more hospitalizations due to acute decompensated heart failure
Mean number of unplanned heart failure hospitalizations | 6 and 12 months
  Mean number of unplanned hospital admissions due to acute decompensated heart failure
Emergency Room visits | 6 and 12 months
  Mean number of emergency room visits
All-cause mortality | 6 and 12 months
  Number of deaths from any cause
Medication adherence - Dose count | 6 and 12 months
  Percentage of prescribed number of doses taken. Assessed throughout the study with the AARDEX MEMS Cap Smart Pill Bottle.
Medication adherence - Dose days | 6 and 12 months
  Percentage of days the correct number of doses were taken. Assessed throughout the study with the AARDEX MEMS Cap Smart Pill Bottle.
Weighing adherence | 6 and 12 months
  Percentage of days patients used the Withings smart scale to measure their weight
Blood pressure monitoring adherence | 6 and 12 months
  Percentage of days patients used the Withings smart blood pressure cuff to measure their blood pressure
Steps | 6 and 12 months
  Mean number of steps per day assessed with a Fitbit activity tracker
Moderate-to-vigorous physical activity (MVPA) minutes | 6 and 12 months
  Average number of MVPA minutes per day assessed with a Fitbit activity tracker
Self-care maintenance | 3, 6, 9, and 12 months
  Mean change in self-care maintenance scores from baseline, assessed with the Self-care Heart Failure Index v 7.2. Scores range from 0 to 100. Higher scores indicate better self-care maintenance.
Symptom perception | 3, 6, 9, and 12 months
  Mean change in symptom perception scores from baseline, assessed with the Self-care Heart Failure Index v 7.2. Scores range from 0 to 100. Higher scores indicate better symptom perception.
Self-care management | 3, 6, 9, and 12 months
  Mean change in self-care management scores from baseline, assessed with the Self-care Heart Failure Index v 7.2. Scores range from 0 to 100. Higher scores indicate better self-care management
Self-care efficacy | 3, 6, 9, and 12 months
  Mean change in self-care efficacy scores from baseline, assessed with the Self-care Heart Failure Index v 7.2. Scores range from 0 to 100. Higher scores indicate better self-care efficacy.
Health Status | 3, 6, 9, and 12 months
  Mean change in health status scores from baseline. Health Status will be assessed with the Kansas City Cardiomyopathy Questionnaire, which contains 23-items that can be quantified into five subscales: physical limitations, symptoms (frequency, severity, and change over time), quality of life (QoL), social interference, and self-efficacy. Lower scores indicate worse health status
Heart Failure Knowledge | 3, 6, 9, and 12 months
  Mean change in heart failure knowledge score from baseline. Assessed with the Dutch Heart Failure Knowledge Questionnaire. Higher scores indicate better knowledge.

CONTACTS AND LOCATIONS:
Overall Officials: Spyros Kitsiou, PhD, Principal Investigator — University of Illinois Chicago
Locations (2):
- United States (2):
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois Hospital & Health Sciences System, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No